CLINICAL TRIAL: NCT04643717
Title: Evaluation of pupillometrY for External Ventricular Drains Stop
Acronym: EYES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/CHU/01
Record Dates: First submitted 2020-11-06; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: All Indication for External Ventricular Drain Clamping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intensive care patients
  Interventions: Other: Electronic pupillometer analysis

INTERVENTIONS:
Other: Electronic pupillometer analysis — Electronic pupillometer analysis

SUMMARY:
Placement of an external ventricular shunt is one of the most common neurosurgical procedures in neuro-resuscitation. However, the modalities of its withdrawal are not, the subject of recommendations but rather of service habits. It has been recently demonstrated that pupillary monitoring by an electronic pupillometer was more reliable than standard clinical monitoring in brain injury patients. This tool provides access to a rich pupillary semiology at the patient's bed.

So the goal is to study the evolution of the various pupillary parameters analyzed by the electronic pupillometer during the external ventricular shunt weaning tests and to highlight the predictive factors of failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients for whom the doctor orders an external ventricular bypass clamp test
* Neuro-injured patients and non-neuro-injured patients whose state of health requires sedation and mechanical ventilation

Exclusion Criteria:

* Ophthalmological pathology making impossible to carry out measurements by the pupillometer (chemosis, eyelid edema, enucleation, etc.).
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have benefited from an external ventricular bypass, whatever the indication, and for whom the doctor in charge prescribes a clamping test.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
The difference in pupillary contraction speed during the photomotor reflex measured by electronic pupillometer as a function of the outcome of the External ventricular lead clamping test | 48 HOURS

SECONDARY OUTCOMES:
Comparison of the pupillometry parameters between neuro wronged's patients and not neuro wronged's patients (parameters measured by pupillometer) | 48 HOURS

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital La Timone, Marseille
  - CHU de la Réunion, Saint-Pierre